CLINICAL TRIAL: NCT01593956
Title: Influence of Anodal Transcranial Direct Current Stimulation on Cortical Plasticity in Concussed Athletes and Healthy Volunteers
Brief Title: Influence of Transcranial Direct Current Stimulation on Cortical Plasticity in Concussed Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Jonathan List, MD, Charite University, Berlin, Germany
Purpose: Treatment
Other Study IDs: EA1/021/12
Record Dates: First submitted 2012-05-07; First posted 2012-05-08 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Concussed Athletes; Healthy Controls
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Concussed athletes (Other)
  Interventions: Behavioral: tDCS
- Healthy controls (Other)
  Interventions: Behavioral: tDCS

INTERVENTIONS:
Behavioral: tDCS

SUMMARY:
Concussed athlethes have discrete decreased abilities in motor learning. Recent research could further show, that cortical plasticity, as measured by transcranial magnetic stimulation (TMS) is reduced. This is possibly due to an increased GABAergic activity, what have been found in concussed athletes by paired pulse protocols in TMS.

GABAergic acitivty can be modulated by transcranial direct current stimulation (tDCS) in a polar-specific manner: anodal tDCS was able to decrease GABA, whereas cathodal tDCS increased tDCS.

Our study aimes to assess the influence of anodal tDCS on cortical plsticity in concussed athlethes. We hypothesize, that anodal tDCS is able to increase cortical plsticity in concussed athlethes.

ELIGIBILITY:
Inclusion Criteria:

* history of at least 2 sports concussion
* age 18 - 50 years

Exclusion Criteria:

* structural deficit on cerebral MRI
* Epilepsy
* neurological disorder
* intake of CNS-active drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Improvement of cortical plasticity after anodal tDCS in concussed athletes

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan List, MD, Principal Investigator — Charité - Department of Neurology; Agnes Flöel, Prof., Principal Investigator — Charité - Department of Neurology
Locations (1):
- Charité - Department of neurology, Berlin, Germany

REFERENCES:
- [Background] De Beaumont L, Tremblay S, Poirier J, Lassonde M, Theoret H. Altered bidirectional plasticity and reduced implicit motor learning in concussed athletes. Cereb Cortex. 2012 Jan;22(1):112-21. doi: 10.1093/cercor/bhr096. Epub 2011 May 13. PMID 21572090
- [Background] Stagg CJ, Bachtiar V, Johansen-Berg H. The role of GABA in human motor learning. Curr Biol. 2011 Mar 22;21(6):480-4. doi: 10.1016/j.cub.2011.01.069. Epub 2011 Mar 3. PMID 21376596
- [Background] Stagg CJ, Best JG, Stephenson MC, O'Shea J, Wylezinska M, Kincses ZT, Morris PG, Matthews PM, Johansen-Berg H. Polarity-sensitive modulation of cortical neurotransmitters by transcranial stimulation. J Neurosci. 2009 Apr 22;29(16):5202-6. doi: 10.1523/JNEUROSCI.4432-08.2009. PMID 19386916